CLINICAL TRIAL: NCT03128775
Title: School Randomized Factorial Trial for Nudging Students Towards Healthy Diet and Physical Activity to Prevent Obesity: a Study Protocol
Brief Title: Nudging Students Towards Healthy Diet and Physical Activity to Prevent Obesity
Acronym: PAAPASNudge
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding was provided by the financial agency
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Oswaldo Cruz Foundation (Other); University of Copenhagen (Other); Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rosely Sichieri, Full professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nudgepaappas
Record Dates: First submitted 2016-10-04; First posted 2017-04-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Primary Prevention

STUDY DESIGN:
Intervention Model Description: PAAPPAS Nudge is a randomized community-based, school-based trial designed to promote healthful choices in a low-income scenario, with will be held in 2018 school-year in 18 municipal public schools in the municipality of Duque de Caxias, metropolitan area of Rio de Janeiro, Brazil (http://duquedecaxias.rj.gov.br/portal/). All students from the 5th and 6th grade from the 18 selected schools will be invited to participate to the study.
  The study design will be of the factorial type, with 4 group arms:
  A) Group 1: control (without any activity); B) Group 2: will receive educational activities in the classroom; C) Group 3: will receive changes in the school environment (nudge strategies); D) Group 4: will receive educational activities and changes in the school environment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nudge (Experimental): This group will receive changes in the school environment (nudge strategies). Interventions regarding food consumption were based on nudge strategies to led students to eat more fruits and vegetables. To stimulate physical activity, several sports equipment (basketball hoops, volleyball nets, balls, ropes, shuttlecock and a lot of toys) are available for use in the school sports court.
  Interventions: Behavioral: Nudge
- Primary prevention (Experimental): This group will receive educational activities in the classroom. Classroom-based educational activities will be based on an earlier study, called PAPPAS, which was developed in the same city and constituted a school-based intervention with the objective of reducing the consumption of sweetened beverages and biscuits and increase the consumption of fruits, vegetables and beans.
  Interventions: Behavioral: Primary prevention
- Primary prevention + nudge (Experimental): This group will receive educational activities and in the classroomchanges in the school environment (nudge).
  Interventions: Behavioral: Primary prevention + nudge
- Control (No Intervention): without any activity

INTERVENTIONS:
Behavioral: Nudge — School lunchrooms are the central place of modifications regarding food consumption, where the following strategies will be conducted:
  1. arrange the fruits served in the school lunch in a prominent position, in containers of bright and contrasting colors to serve them;
  2. Create creative names for food served at meals will be created by the students used on displays at canteen tables, posters on the way of the cafeteria and at a menu outside the cafeteria.
  To encourage water consumption, footprints that lead to them to water fountains will be painted on the floor. To stimulate physical activity, several sports equipment (basketball hoops, volleyball nets, balls, ropes, shuttlecock and a lot of toys) will be available for use in the school sports court. The courts will be renovated and footsteps painted in order to nudging students to the sports equipment.
  Arms: Nudge
Behavioral: Primary prevention — Classroom-based educational activities based on an earlier study, called PAPPAS, which was developed in the same city and constituted a school-based intervention with the objective of reducing the consumption of sweetened beverages and biscuits and increase the consumption of fruits, vegetables and beans. Activities will be facilitated by trained research assistants. Printed instructions and orientations on the facilitation process will support the assistants' efforts. The activities will require 20 to 30 minutes, and teachers will be encouraged to reiterate the message during their lesson. The goal is to promote ten one-hour sessions of activity for each class.
  Arms: Primary prevention
Behavioral: Primary prevention + nudge — This group will receive both primary prevention and nudge activities. At school lunchrooms, the fruits served in the school lunch will be put in a prominent position, in containers of bright and contrasting colors to serve them; create creative names for food served at meals will be created by the studentes, footprints that lead to them to water fountains will be painted on the floor. Several sports equipment (basketball hoops, volleyball nets, balls, ropes, shuttlecock and a lot of toys) will be available for use in the schools sport court. Also, classroom-based educational activities based on an earlier study, called PAPPAS, will be held. The activities will require 20 to 30 minutes, and teachers will be encouraged to reiterate the message during their lesson. The goal is to promote ten one-hour sessions of activity for each class.
  Arms: Primary prevention + nudge

SUMMARY:
The objective of the present study is to estimate the effect of nudging proposals on the students' Body Mass Index, based on changes made in the school environment. This is a factorial randomized community trial, which will be conducted in 18 public schools in the city of Duque de Caxias, RJ.

ELIGIBILITY:
Inclusion Criteria:

5th and 6th grades students consent form signed by parents/tutors

Exclusion Criteria:

pregnant girls

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body mass Index (BMI) | 1 year
  The body weight will be measured by a portable electronic scale with a segmental body composition monitor (Tanita BC-558). The height will be measure by a portable stadiometer (brand: "AlturaExata"). BMI will be calculated as weight/stature*stature.

SECONDARY OUTCOMES:
body fat percentage | 1 year
  Body fat percentage will be measured by a portable electronic scale with a segmental body composition monitor (Tanita BC-558).

CONTACTS AND LOCATIONS:
Locations (1):
- 18 Schools of Metropolitan Area, Duque de Caxias, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No